CLINICAL TRIAL: NCT06195787
Title: Assessing the Safety and Efficiency of a Simplified Diagnostic Approach for Deep Vein Thrombosis
Brief Title: Improving Emergency Department Testing for Deep Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Dr. Kerstin de Wit (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Sponsor-Investigator, Dr. Kerstin de Wit, Associate Professor Department of Emergency Medicine, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 3717
Record Dates: First submitted 2023-12-18; First posted 2024-01-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Deep Vein Thrombosis (DVT)
Keywords: deep vein thrombosis; venous thromboembolism; emergency medical services; diagnosis
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study will use a new way to test for deep vein thrombosis (DVT) of the leg. A DVT is a blood clot in the leg and is a medical problem that can cause swelling, pain, and redness. If the blood clot is not treated, it can cause more serious, long-term effects, and occasionally lead to death.

The main questions the study aims to answer are:

1. How safe is our new blood clot testing method?
2. How efficient is our new blood clot testing method?

The study will be run in the emergency department and urgent care centre in Kingston, Ontario. Patients who are tested for a DVT in the leg can be included in the study. Researchers follow the patient through chart review to make sure the new system is safe and efficient.

ELIGIBILITY:
Inclusion Criteria:

- emergency physician decides to test for DVT of the lower limb.

Exclusion Criteria:

* <18 years of age;
* tested for DVT without using the ToDay algorithm at the index visit;
* D-dimer level is known before ToDay item assessment;
* a new indication for anticoagulation at the emergency department assessment (other than DVT) in a patient not previously prescribed an anticoagulant;
* a history of prior lower limb DVT, where there is no access to baseline ultrasound imaging;
* suspected of having a pulmonary embolism;
* has previously participated in this study;
* has previously opted out of all research at hospital site;
* left the emergency department or urgent care centre against medical advice;
* D-dimer was ordered prior to initial physician assessment;
* imaging for DVT or pulmonary embolism within the previous 30 days;
* transferred from another hospital organization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be enrolled after a visit to the Kingston Health Sciences emergency department and urgent care centre in Kingston, Ontario.
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
False negative rate of the new DVT testing | This will be measured at 30-days after the patient's index emergency department visit.
  This is the proportion of patients who have DVT excluded by the new ToDay protocol and who were subsequently diagnosed with either a lower limb DVT or pulmonary embolism.

SECONDARY OUTCOMES:
Efficiency of the new DVT testing | At the index emergency department visit.
  This is the proportion of all study patients who do not require ultrasound imaging at index visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No